CLINICAL TRIAL: NCT01917656
Title: Efficacy and Safety of Liraglutide Versus Sulphonylurea Both in Combination With Metformin During Ramadan in Subjects With Type 2 Diabetes
Acronym: LIRA-Ramadan™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-3987; U1111-1132-9716 (Other: WHO)
Record Dates: First submitted 2013-07-29; First posted 2013-08-07 (Estimated); Results first posted 2015-10-07 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide+Metformin (Experimental): Liraglutide 1.8 mg administered once daily subcutaneously, in combination with pre-trial tablet metformin of unchanged dose.
  Interventions: Drug: liraglutide; Drug: metformin
- Sulphonylurea and Metformin (Active Comparator): Subjects continued on pre-trial sulphonylurea tablet treatment, in combination with pre-trial tablet metformin of unchanged dose.
  Interventions: Drug: metformin; Drug: sulphonylurea

INTERVENTIONS:
Drug: liraglutide — 1.8 mg administered subcutaneously (s.c., under the skin) once daily
  Arms: Liraglutide+Metformin
Drug: metformin — Subjects will continue on their pre-trial metformin tablet treatment, dose unchanged
Drug: sulphonylurea — Subjects will continue on their pre-trial SU tablet treatment, doses unchanged
  Arms: Sulphonylurea and Metformin

SUMMARY:
This trial is conducted in Africa and Asia. The aim of the trial is to investigate the efficacy and safety of liraglutide versus sulphonylurea (SU) both in combination with metformin during Ramadan in subjects with type 2 diabetes (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* - Subjects diagnosed with T2DM and treated with metformin equal to or above 1000 mg/day and SU (gliclazide, glipizide or glyburide/glibenclamide at maximum tolerated dose (at least half maximum approved dose) or glimepiride at maximum tolerated dose (at least 2 mg/day)), both at a stable dose for at least 90 days prior to screening. Stable is defined as unchanged medication and dose
* - HbA1c 7.0-10.0% (53- 86 mmol/mol) (both inclusive)
* - Body Mass Index (BMI) equal to or above 20 kg/m^2
* - Subjects who have expressed their intention to fast (daytime, i.e. between sunrise and sunset) during Ramadan after receiving medical counselling regarding the risk of fasting

Exclusion Criteria:

* - Any contraindication for successful and sustained fasting from a medical perspective at the discretion of the investigator (such as acute illness, severe hypoglycaemia within 90 days prior to screening, a history of recurrent hypoglycaemia, hypoglycaemia unawareness, ketoacidosis within 90 days prior to screening, hyperosmolar hyperglycaemic coma within 90 days prior to screening, subjects performing intense physical labour)
* - Any chronic disorder or severe disease which, in the opinion of the investigator might jeopardise subject's safety or compliance with the protocol
* - History of chronic pancreatitis or idiopathic acute pancreatitis
* - Screening calcitonin value equal to or above 50 ng/L
* - Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2)
* - Impaired liver function, defined as alanine aminotransferase (ALAT) equal to or above 2.5 times upper normal limit (UNL)
* - Impaired renal function defined as estimated glomerular filtration rate (eGFR) below 60 mL/min/1.73 m^2 per Modification of Diet in Renal Disease (MDRD) formula)
* - Any episode of unstable angina, acute coronary event, cerebral stroke/transient ischemic attack (TIA) or other significant cardiovascular event as judged by the investigator within 90 days prior to screening
* - Diagnosis of malignant neoplasm in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2014-01-09 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2014-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (33):
- Algeria (5):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Constantine
  - Novo Nordisk Investigational Site, Oran
  - Novo Nordisk Investigational Site, Sétif
  - Novo Nordisk Investigational Site, Sidi Bel Abbes
- India (6):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mysore, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
- Israel (3):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
- Lebanon (2):
  - Novo Nordisk Investigational Site, Beirut
  - Novo Nordisk Investigational Site, Lebanon - Beirut
- Malaysia (7):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Ipoh, Perak
  - Novo Nordisk Investigational Site, Klang, Selangor
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Putrajaya
  - Novo Nordisk Investigational Site, Selangor Darul Ehsan
  - Novo Nordisk Investigational Site, Seremban, Negeri Sembilan
- South Africa (5):
  - Novo Nordisk Investigational Site, Benoni, Gauteng
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Lenasia, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
- United Arab Emirates (5):
  - Novo Nordisk Investigational Site, Ajman
  - Novo Nordisk Investigational Site, Dubai
  - Novo Nordisk Investigational Site, Ras al-Khaimah
  - Novo Nordisk Investigational Site, Sharjah city
  - Novo Nordisk Investigational Site, Umm Al Quwain City

REFERENCES:
- [Result] Azar ST, Echtay A, Wan Bebakar WM, Al Araj S, Berrah A, Omar M, Mutha A, Tornoe K, Kaltoft MS, Shehadeh N. Efficacy and safety of liraglutide compared to sulphonylurea during Ramadan in patients with type 2 diabetes (LIRA-Ramadan): a randomized trial. Diabetes Obes Metab. 2016 Oct;18(10):1025-33. doi: 10.1111/dom.12733. Epub 2016 Aug 18. PMID 27376711
- [Derived] Lee SWH, Chen WS, Sellappans R, Md Sharif SB, Metzendorf MI, Lai NM. Interventions for people with type 2 diabetes mellitus fasting during Ramadan. Cochrane Database Syst Rev. 2023 Jul 12;7(7):CD013178. doi: 10.1002/14651858.CD013178.pub2. PMID 37435938
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 39 sites in 7 countries as follows: Algeria: 7 sites; Israel: 4 sites; India: 5 sites; Lebanon: 2 sites; Malaysia: 7 sites; South Africa: 8 sites; United Arab Emirates: 6 sites
Pre-assignment Details: Subjects were randomised in a 1:1 manner to either switch to liraglutide 1.8 mg/day added on to metformin or to continue their pre-trial SU and metformin treatment.
Groups:
- Liraglutide and Metformin: Liraglutide 1.8 mg administered once daily subcutaneously, in combination with pre-trial tablet metformin of unchanged dose.
- Sulfonylurea and Metformin: Subjects continued on pre-trial sulfonylurea tablet treatment, in combination with pre-trial tablet metformin of unchanged dose.
Period: Overall Study
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Started | 172 | 171
Exposed | 171 (1 subject was withdrawn prior to exposure to trial products) | 170 (1 subject was withdrawn prior to exposure to first SU dose after randomisation)
Exposed During Ramadan (Fasting) | 152 | 163
Completed | 146 | 147
Not Completed | 26 | 24
Not completed — Adverse Event | 11 | 0
Not completed — Withdrawal criteria | 8 | 14
Not completed — Unclassified | 0 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin | Total
Number analyzed (Participants) | 171 | 170 | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (9.27) | 54.0 (9.33) | 54.5 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 87 | 173
  Male | 85 | 83 | 168

OUTCOME MEASURES:

1. Primary Outcome: Change in Fructosamine From Start of Ramadan to End of Ramadan
Description: The level of fructosamine in the blood was used to assess the glycaemic control in the patients during the time period described- from start of Ramadan (day -1, visit 8) to end of Ramadan (day 29, visit 12).
Time Frame: Day -1, day 29
Population: Full analysis set (FAS). The number of subjects in FAS were 171 (Liraglutide) and 169 (Sulfonylurea), few subjects did not contribute to this analysis.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Number analyzed (Participants) | 146 | 151
umol/L | -13.2 (36.0) | -14.9 (43.0)

2. Secondary Outcome: Fructosamine at End of Ramadan
Description: The fructosamine values at the end of Ramadan (visit 12) were presented
Time Frame: Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Number analyzed (Participants) | 146 | 151
umol/L | 276.8 (44.1) | 284.9 (46.6)

3. Secondary Outcome: Change From Start of Ramadan to End of Ramadan in Fasting Plasma Glucose (FPG)
Description: The level of FPG in the blood of fasting patients was addressed to monitor glycaemic control during the period described.
Time Frame: Day -1, day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Number analyzed (Participants) | 146 | 157
mmol/L | -0.1 (2.0) | 0.1 (3.8)

4. Secondary Outcome: Change From Baseline to End of Ramadan in Fasting Plasma Glucose
Description: The changes from baseline measured postbaseline (i.e., the changes measured on visit 8 and 12) entered as the dependent variables, and visit, treatment, country, and the stratification variables were included as fixed factors and the corresponding values for the specific endpoint measured at randomisation as covariate.
Time Frame: Baseline, day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Number analyzed (Participants) | 143 | 156
mmol/L | -1.8 (3.1) | -0.6 (3.6)

5. Secondary Outcome: Change From Baseline to End of Ramadan in Glycosylated Haemoglobin (HbA1c)
Description: The level of glycosylated haemoglobin in blood was used to assess the glycaemic control of the patients during the time period described.
Time Frame: Baseline, day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Number analyzed (Participants) | 146 | 156
Percent (%) glycosylated haemoglobin | -1.3 (1.1) | -0.7 (0.9)

6. Secondary Outcome: Change From Baseline to End of Ramadan in Body Weight
Time Frame: Baseline, day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Number analyzed (Participants) | 165 | 168
kg | -5.40 (0.2205) | -1.46 (0.2139)

7. Secondary Outcome: Subjects Who at End of Treatment (4 Weeks Post Ramadan) Achieve (y/n): HbA1c Below 7.0% (53 mmol/Mol) (ADA Target)
Description: Subjects who at end of treatment (Visit 14, 4 weeks post Ramadan) achieve (y/n): HbA1c below 7.0% (53 mmol/mol) (ADA target)
Time Frame: Visit 14 (4 weeks post Ramadan)
Population: Full analysis set
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Number analyzed (Participants) | 171 | 169
percentage (%) of subjects | 51.0 | 29.9

8. Secondary Outcome: Subjects Who at End of Treatment (4 Weeks Post Ramadan) Achieve (y/n): HbA1c Below 7.0% (53 mmol/Mol), and no Confirmed Hypoglycaemic Episodes
Description: as for outcome 7
Time Frame: Visit 14 (4 weeks post Ramadan)
Population: Full analysis set
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Number analyzed (Participants) | 171 | 169
percentage (%) of subjects | 47.6 | 25.2

9. Secondary Outcome: Number of Confirmed Hypoglycaemic Episodes During Ramadan (Fasting), Based on Each Subject's Individual Fasting Period.
Time Frame: Day -1 to day 29
Population: Safety analysis set
Measure: Number; unit: Events/1000 years of patient exposure
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Number analyzed (Participants) | 152 | 163
Events/1000 years of patient exposure | 246 | 623

10. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) During Ramadan (Fasting), Based on Each Subject's Individual Fasting Period.
Description: A serious AE was an experience that at any dose resulted in any of the following: Death, a life-threatening experience, in-patient hospitalisation or prolongation of existing hospitalisation, a persistent or significant disability or incapacity, congenital anomaly or birth defect, important medical events.
  Mild - no or transient symptoms, no interference with the subject's daily activities Moderate - marked symptoms, moderate interference with the subject's daily activities Severe - considerable interference with the subject's daily activities, unacceptable
Time Frame: Day -1 to day 29
Population: Safety analysis set
Measure: Number; unit: Events/1000 years of patient exposure
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Number analyzed (Participants) | 152 | 163
Events/1000 years of patient exposure
  Adverse events | 5258 | 3349
  Serious adverse events | 164 | 0
  Severe adverse events | 411 | 78
  Moderate adverse event | 986 | 779
  Mild adverse event | 3861 | 2492

ADVERSE EVENTS:
Time Frame: A treatment emergent AE during Ramadan (fasting) had onset on or after the individual subject's first day of Ramadan fasting, and no later than the individual subject's last day of Ramadan fasting.
Description: Safety analysis set included all randomised subjects who were exposed to the trial drug. Subjects in the safety analysis set contributed to the evaluation 'as treated'. A total of 315 randomised subjects were exposed to trial products during Ramadan (fasting), of which 152 subjects were exposed to liraglutide and 163 subjects were exposed to SU.
Arm/Group | Liraglutide and Metformin | Sulfonylurea and Metformin
Serious Adverse Events (participants affected / at risk) | 2/152 | 0/163
Other Adverse Events (participants affected / at risk) | 8/152 | 1/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide and Metformin (N=152) | Sulfonylurea and Metformin (N=163)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide and Metformin (N=152) | Sulfonylurea and Metformin (N=163)
Vomiting (Gastrointestinal disorders) | 8 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.